CLINICAL TRIAL: NCT02333747
Title: The Effects of Transcutaneous Electrical Acupoint Stimulation on the Quality of Recovery After Thyroidectomy Surgery
Brief Title: Can Transcutaneous Electrical Acupoint Stimulation Improve the Quality of Recovery After Thyroidectomy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K2014-12-003
Record Dates: First submitted 2015-01-02; First posted 2015-01-07 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2015-07

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the TEAS group (Experimental): Patients in the TEAS group received pre-operative TEAS for 30 min before the induction of anesthesia using the Hans electronic acupuncture apparatus (HANS-100A, Nanjing Jisheng Medical Technology Company, Nanjing, China) in the holding area. TEAS was applied to two pairs of acupoints: bilateral Hegu (LI4) and Neiguan (PC6).
  Interventions: Device: the Hans electronic acupuncture apparatus
- the sham group (Sham Comparator): In the sham group, the patients were connected to the Hans electronic acupuncture apparatus (HANS-100A, Nanjing Jisheng Medical Technology Company, Nanjing, China), but electronic stimulation was not applied.
  Interventions: Device: the Hans electronic acupuncture apparatus

INTERVENTIONS:
Device: the Hans electronic acupuncture apparatus — TEAS was performed with a dense-disperse frequency of 2/10 Hz and an intensity of 6-9 mA for 30 min using the Hans electronic acupuncture apparatus (HANS-100A, Nanjing Jisheng Medical Technology Company, Nanjing, China).

SUMMARY:
The effect of transcutaneous electric acupoint stimulation (TEAS) on the quality of recovery in patients undergoing thyroidectomy surgery remains unclear. Therefore, the investigators conducted this prospective, randomized, double-blind study to verify the hypothesis that pre-operative TEAS could improve the quality of recovery (QoR) after thyroidectomy surgery.

DETAILED DESCRIPTION:
Transcutaneous electric acupoint stimulation (TEAS) is a form of non-invasive electrical stimulation that produces a perceptible sensation via electrodes attached to the skin. It has no risk of infections and can potentially be applied by medical personnel with minimal training. Clinical trials have demonstrated that TEAS reduces the consumption of intra-operative anesthetics and general anesthesia related side-effects.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive female patients aged 18 to 60 with American Society of Anesthesiologists physical status (ASA) physical status I or II, who underwent general anesthesia for elective thyroidectomy surgery

Exclusion Criteria:

* potentially difficult airway,
* a history of chronic pain,
* drug or alcohol abuse,
* mental disorder,
* intake of any analgesic drug within 48 h before surgery, and
* previous experience with acupuncture treatment

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
the quality of recovery, as measured by a 40-item questionnaire | 24 hours after surgery
  The primary outcome was the quality of recovery, which was assessed on the day before surgery and 24 h after surgery using a 40-item questionnaire (QoR-40)

SECONDARY OUTCOMES:
the incidence of postoperative nausea and vomiting | 24 hours after surgery
postoperative pain intensity, as assessed using Visual Analogue Scale (VAS) | 24 hours after surgery
patient's satisfaction, as evaluated with a 10-point numerical rating scale: 10= excellent, 1= bad. | at 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Chen, MD, Study Director — Fujian Provincial Hospital, China
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen Y, Yang Y, Yao Y, Dai D, Qian B, Liu P. Does transcutaneous electric acupoint stimulation improve the quality of recovery after thyroidectomy? A prospective randomized controlled trial. Int J Clin Exp Med. 2015 Aug 15;8(8):13622-7. eCollection 2015. PMID 26550304